CLINICAL TRIAL: NCT04494581
Title: Assessment of Practices and of Immunization Programs Against Flu and Pertussis in Maternity Hospitals
Brief Title: GriCoVax Study in 4 Maternity Wards in the Ile-de-France Region
Acronym: GriCoVax
Status: Completed | Type: Observational
Sponsor: Groupe d'Etude sur le Risque d'Exposition des Soignants aux Agents Infectieux (Network)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government); National Agency of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: GriCoVax - GERES; 2019-A00346-51 (Other: ANSM)
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Pertussis Vaccine; Healthcare Worker Patient Transmission; Pregnant Women; Influenza Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant and postpartum women: Pregnant and postpartum women over 18, meeting inclusion and exclusion criteria.
  Interventions: Other: questionnaire
- healthcare workers: Health professionals over 18, working in maternity wards included.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Questionnaire survey

SUMMARY:
Implementation of organizational adjustments can enhance involvement of healthcare teams in carrying out flu and pertussis vaccinations, and optimizing access to vaccines for women and their families. Pertussis vaccination of pregnant women is envisaged by the French Health Autority, considering that, given international experiences, vaccination during the second trimester of pregnancy is safe, effective, and would aim to protect babies during the first months of their life. Before considering such a recommendation in France, the acceptability of this strategy by pregnant women and health professionals must be considered.

DETAILED DESCRIPTION:
Multicentre, descriptive study conducted in a declarative manner and supplemented by direct observation by an investigator.

Main objectives:

* Assess existing practices of the various actors involved in flu and pertussis vaccination of pregnant or postpartum women medically followed in maternity wards.
* Assess acceptability of pertussis and flu vaccination during pregnancy by women medically followed in maternity wards, and by health professionals of theses facilities.

Secondary objectives:

* Assess flu and pertussis immunization coverage of pregnant and postpartum women and of health professionals working in maternity wards.
* Assess the links between immunization coverage of health professionals and their current practices in promoting flu and pertussis vaccination of women in maternity wards.

Main outcome measures:

* Identify in each maternity hospital facilitators of flu and pertussis vaccination.
* Proportion of women willing to be vaccinated against pertussis and flu during pregnancy.
* Proportion of health professionals agreeing to vaccinate pregnant women against flu and pertussis.

Secondary endpoints:

* Flu and pertussis immunization coverage of pregnant and postpartum women.
* Flu and pertussis immunization coverage of health professionals.
* Proportion of patient records with vaccination trace.
* Link between understanding of vaccines and vaccine-preventable diseases, and immunization coverage of health professionals.
* Link between attitudes and practices of health professionals, and immunization coverage of patients.
* Link between immunization coverage of patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

Pregnant and postpartum women over 18 medically followed in maternity wards included. Femmes enceintes ou en post-partum :

Health professionals over 18 working in maternity wards included.

Exclusion Criteria:

Women under the protection of a conservator Temporary Health staff

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer women and staff.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Identify in each maternity hospital facilitators of flu and pertussis vaccination | May 2019 - July 2019
  Qualitative interviews
Proportion of women willing to be vaccinated against pertussis and flu during pregnancy | September 2019-December 2019
  Questionnaire survey
Proportion of health professionals agreeing to vaccinate pregnant women against flu and pertussis. | October 2019-February 2020
  Questionnaire survey

SECONDARY OUTCOMES:
Flu and pertussis immunization coverage of pregnant and postpartum women | September 2019-December 2019
  Questionnaire survey
Flu and pertussis immunization coverage of health professionals | October 2019-February 2020
  Two survey Questionnaires: one distributed to health professionals, one addressed to Occupational Health services
Proportion of patient records with vaccination trace | October-December 2019
  Review of sample of patient records

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Maternité Hôpital privé, Antony
  - Maternité Hôpital Jean Verdier, Bondy
  - Maternité Notre Dame de Bon Secours - GH Paris St Joseph, Paris
  - Maternité Port Royal, Paris

IPD SHARING:
Plan to Share IPD: No